CLINICAL TRIAL: NCT04460053
Title: A Prospective Feasibility Trial Measuring Neurofilament Light Protein in Peripheral Blood as a Biomarker for Neurotoxicity After Isolated Limb Perfusion.
Brief Title: Neurofilament Light Protein in Peripheral Blood Used as a Biomarker for Neurotoxicity After Isolated Limb Perfusion.
Acronym: ILP-NfL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Principal Investigator, Roger Olofsson Bagge, Associate professor, Vastra Gotaland Region
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ILP-NfL
Record Dates: First submitted 2019-05-09; First posted 2020-07-07 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Malignant Melanoma
Keywords: toxicity; biomarker; Neurofilament Light protein; In-transit metastasis; Hyperthermic isolated limb perfusion
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: A prospective feasibility trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurofilament light protein measurement (Experimental): Neurofilament light protein measurements in peripheral blood pre- peri- and postoperatively.
  Interventions: Procedure: Neurofilament light protein measurement in Isolated limb perfused patients

INTERVENTIONS:
Procedure: Neurofilament light protein measurement in Isolated limb perfused patients — A prospective feasibility trial measuring neurofilament light protein in peripheral blood as a biomarker for neurotoxicity after isolated limb perfusion.

SUMMARY:
A prospective feasibility trial initially including 10 patients to investigate if Neurofilament light protein can be detected in peripheral blood in patients undergoing Isolated Limb Perfusion with chemotherapeutic agents. This biomarker could act as predictive biomarker for neurotoxicity after isolated limb perfusion.

DETAILED DESCRIPTION:
In isolated limb perfusion (ILP) neurotoxicity is a known side effect, this is in spite of the fact that a relatively mild hyperthermic temperature is used which should be well tolerated by the nerves and other normal tissues in the limbs. It seems probable that the neurotoxicity observed after ILP results from both a thermal enhancement of drug toxicity combined with a local effect of a high tourniquet pressure that is used to isolate the blood flow. Prevention of regional and systemic toxicity is essential for improving the outcome after the procedure. It is known that both higher doses of melphalan, higher temperatures and longer perfusion time correlates to a higher toxicity. The Wieberdink method is a grading system for the reaction of the normal tissues after ILP and the grading is used as a routine in ILP today. Neurofilament light protein (NfL) is released into the cerebrospinal fluid (CSF) during axonal damage and has been shown to be elevated in different forms of dementia. An NfL assay sensitive enough to measure NfL in blood was recently developed. Its concentration reflects axonal injury in both central and peripheral nervous system disorders.The primary aim of this study is to investigate the possibility to measure neurofilament as a biomarker for peripheral nerve toxicity after isolated limb perfusion.

ELIGIBILITY:
Inclusion Criteria:

1. Patient scheduled for treatment with isolated limb perfusion
2. Age over 18 years
3. Signed informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-04-12 (Actual); Primary Completion 2020-09-18 (Actual); Study Completion 2020-10-25 (Actual)

PRIMARY OUTCOMES:
Neurofilament light protein measurement in peripheral blood | 1 day postoperatively
  Neurofilament light protein
Neurofilament light protein measurement in peripheral blood | 3 days postoperatively
  Neurofilament light protein
Neurofilament light protein measurement in peripheral blood | 4 weeks postoperatively
  Neurofilament light protein

CONTACTS AND LOCATIONS:
Overall Officials: Roger Olofsson Bagge, Principal Investigator — Sahlgrenska University Hospital, Department of Sugery
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Corderfeldt Keiller A, Axelsson M, Bragadottir G, Blennow K, Zetterberg H, Olofsson Bagge R. A prospective feasibility trial exploring novel biomarkers for neurotoxicity after isolated limb perfusion. Perfusion. 2024 Nov;39(8):1657-1666. doi: 10.1177/02676591231213506. Epub 2023 Nov 7. PMID 37933726
- [Derived] Corderfeldt Keiller A, Holmen A, Hansson C, Ricksten SE, Bragadottir G, Olofsson Bagge R. Non-invasive and invasive measurement of skeletal muscular oxygenation during isolated limb perfusion. Perfusion. 2023 Jul;38(5):1019-1028. doi: 10.1177/02676591221093201. Epub 2022 May 16. PMID 35575302